CLINICAL TRIAL: NCT02698631
Title: Isolation of Pulmonary Veins With the Aid of Magnetic Resonance Imaging
Acronym: ALICIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); University of Barcelona (Other)
Responsible Party: Principal Investigator, Josep Lluis Mont Girbau, MD PhD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALICIA-FA
Record Dates: First submitted 2016-02-04; First posted 2016-03-04 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Atrial Fibrillation
Keywords: Catheter Ablation; Radiofrequency; Fibrosis; Late-gadolinium enhanced MRI
MeSH Terms: conditions — Atrial Fibrillation; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional AF ablation. (Active Comparator): A standard radiofrequency AF ablation procedure will be carried out without LGE information.
  Interventions: Procedure: Conventional AF ablation
- LGE-MRI guided AF ablation. (Experimental): Fibrosis information obtained from post-processed LGE-MRI will be used to guide AF ablation procedures.
  Interventions: Procedure: LGE-MRI guided AF ablation

INTERVENTIONS:
Procedure: Conventional AF ablation — Conventional AF ablation will be carried out according to the standard procedure. Atrial anatomical MRI information will be integrated into the navigation system. Ablation procedure will be carried out with a Smart Touch® catheter (temperature 45 °C, 40W or 30W for anterior or posterior wall, respectively).
  Both in first and re-do procedures, procedure endpoint will be electrical isolation of all pulmonary veins.
  Arms: Conventional AF ablation.
Procedure: LGE-MRI guided AF ablation — Post-processed LGE-MRI will be used to identify left atrial fibrotic patches and lesions surrounding pulmonary veins (re-do procedures). Both MRI atrial anatomical and fibrosis information will be integrated into the navigation system. Ablation procedures will be carried out with a SmartTouch® catheter (temperature 45°C, 40W or 30W for anterior or posterior wall, respectively).
  * Procedural end-point for first ablation procedures will be isolation of all pulmonary veins, and encirclement and isolation of all atrial fibrotic areas.
  * In re-do procedures, all left atrial fibrosis patches will be encircled and isolated and, for electrically non-isolated pulmonary veins, all anatomical gaps in lesions surrounding pulmonary veins (as identified in LGE-MRI) will be closed.
  Arms: LGE-MRI guided AF ablation.

SUMMARY:
The ALICIA-FA study will elucidate whether targeting atrial myocardial fibrosis identified by late gadolinium-enhanced magnetic resonance imaging (LGE-MRI) improves atrial fibrillation (AF) ablation outcomes.

DETAILED DESCRIPTION:
Atrial fibrosis is a hallmark of the AF substrate. An accurate identification and localization of myocardial fibrosis areas prior to an ablation procedure by means of LGE-MRI might help to target atrial areas harboring AF, thereby improving ablation outcomes and reducing AF recurrences.

In order to test this hypothesis, we will conduct a randomized study comparing the isolation of pulmonary veins without fibrosis imaging (conventional ablation procedure) vs. isolation of the pulmonary veins and pathological (fibrotic) tissue with the aid of LGE-MRI. Fibrotic tissue patches will be encircled and isolated in all patients in the active arm; furthermore, LGE-MRI will be used to identify, locate and guide ablation catheter to anatomical gaps surrounding pulmonary veins in re-do procedures.

Eventually, we will identify an optimized ablation strategy in patients undergoing AF radiofrequency ablation on the basis of left atrium (LA) fibrosis characterization.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a first or subsequent ablation procedure.
* Pre-procedural 3 Tesla LGE-MRI.
* Referred for radiofrequency ablation of pulmonary veins (paroxysmal, persistent or long-standing AF).
* Signed informed consent.

Exclusion Criteria:

* Claustrophobia.
* Refusal to participate in the study.
* Presence of atrial thrombus.
* LA anteroposterior diameter >55 mm.
* Major renal impairment.
* Contrast allergy.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-06 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial arrhythmias, lasting more than 30 sec. | 1 year
  Recurrence is defined as any documented episode of AF/atrial tachycardia lasting more than 30 seconds, after a blanking period of 3 months.

SECONDARY OUTCOMES:
Total time of radiofrequency application | During procedure
Total X-ray time | During procedure

CONTACTS AND LOCATIONS:
Overall Officials: Lluís Mont, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (2):
- Spain (2):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospial Clinic of Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bisbal F, Benito E, Teis A, Alarcon F, Sarrias A, Caixal G, Villuendas R, Garre P, Soto N, Cozzari J, Guasch E, Junca G, Prat-Gonzalez S, Perea RJ, Bazan V, Tolosana JM, Arbelo E, Bayes-Genis A, Mont L. Magnetic Resonance Imaging-Guided Fibrosis Ablation for the Treatment of Atrial Fibrillation: The ALICIA Trial. Circ Arrhythm Electrophysiol. 2020 Nov;13(11):e008707. doi: 10.1161/CIRCEP.120.008707. Epub 2020 Oct 8. PMID 33031713